CLINICAL TRIAL: NCT01653665
Title: Does GM-CSF Restore Effective Neutrophil Function in Critically Ill Patients?
Brief Title: Does GM-CSF Restore Neutrophil Phagocytosis in Critical Illness?
Acronym: GMCSF
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: Medical Research Council (Other Government); Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: AJSEB001; G1100233 (Other Grant/Funding Number: Medical Research Council); 2011-005815-10 (EudraCT Number); ISRCTN95325384 (Other: ISRCTN)
Record Dates: First submitted 2012-07-16; First posted 2012-07-31 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Critical Illness; Sepsis; Immuno-suppression
MeSH Terms: conditions — Critical Illness; Sepsis | interventions — sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Leukine (Sargramostim, GM-CSF) (Active Comparator): Participants in dose finding study will receive either 3 or 6 micrograms per kilo per day as a daily subcutaneous injection for either 4 or 7 days. Within the Randomised controlled trial, participants will receive the dose as chosen following the dose finding study.
  Interventions: Drug: Leukine
- Placebo (normal saline) (Placebo Comparator): Participants in the randomised controlled trial may be randomised to receive a daily subcutaneous injection of normal saline (placebo) for 4 or 7 days as decided following the results of the dose finding study
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Leukine — Daily subcutaneous injection of either 3 or 6 micrograms per kilo per day, for either 4 or 7 days.
  Other Names: Sargramostim; GM-CSF
  Arms: Leukine (Sargramostim, GM-CSF)
Drug: Normal Saline — Patients in the randomised controlled trial may receive this placebo as a single daily subcutaneous injection. The volume will match that of the active drug.
  Other Names: placebo
  Arms: Placebo (normal saline)

SUMMARY:
Despite the introduction of multiple preventative measures rates of hospital acquired infection in the intensive care unit remain high. New approaches to tackling this problem are required. The neutrophil (a type of white blood cell) is the key cell fighting bacterial and fungal infection in the body. This research group has already shown that the majority of patients on intensive care have neutrophils which don't ingest germs effectively and are therefore less able to fight infection. These patients, whose white blood cells don't work properly, are much more likely to develop a second infection whilst in hospital (hospital acquired infection).

Previous work done by this group has shown that by adding a drug called granulocyte macrophagecolony stimulating

factor (GM-CSF) to a sample of blood from these patients in the lab, it is possible to restore the ability of the white blood cells to ingest bacteria and fight infection.

This study will test whether it is possible to restore the capacity of patients' white blood cells to eat germs by giving them GM-CSF as an injection while they are on intensive care.

The study will involve identifying adult patients on intensive care whose white blood cells don't work properly in this way. Patients taking part in the study will receive an injection, under the skin, of either the drug, GM-CSF, or a solution which will have no effect (placebo). The investigators will compare whether those patients who have received the GM-CSF injection have an improvement in the function of the white blood cells compared to those who don't.

As well as looking at the function of the white blood cells the investigators will also study whether there is a difference in the rates of infection picked up in hospital between the two groups.

This study is funded by the Medical Research Council.

ELIGIBILITY:
Inclusion Criteria:

* Fulfil criteria for systemic inflammatory response syndrome on admission to ICU (see appendix 1)
* Has required support of one or more organ systems (invasive ventilation, inotropes or haemofiltration) during current ICU stay
* Survival over next 48 hours deemed most likely outcome by responsible ICU clinician
* Admitted to ICU within last 72 hours
* Neutrophil phagocytic capacity <50%

Exclusion Criteria:

* Absence/refusal of informed consent
* Current prescription of a colony stimulating factor
* Any history of allergy/adverse reaction to GM-CSF
* Total white cell count >30x109/litre at time of screening
* Haemoglobin < 7.5g/dl at the time of screening
* Age < 18 years
* Pregnancy or lactation
* Known in-born errors of neutrophil metabolism
* Known haematological malignancy and/or known to have >10% peripheral blood blast cells
* Known aplastic anaemia or pancytopaenia
* Platelet count <50x109/litre
* Chemotherapy or radiotherapy within the last 24 hours
* Solid organ or bone marrow transplantation
* Use of maintenance immunosuppressive drugs other than maintenance corticosteroids (allowed up to 10mg prednisolone/day or equivalent)
* Known HIV infection
* Active connective tissue disease (e.g. rheumatoid disease, systemic lupus erythematosus) requiring active pharmacological treatment.
* ST-segment elevation myocardial infarction, acute pericarditis (by ECG criteria) or pulmonary embolism (radiographically confirmed) in previous week
* Involvement in any study involving an investigational medicinal product in the previous 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-08; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Neutrophil phagocytosis | 2 days after GMCSF/placebo administration
  neutrophil phagocytic capacity will be measured as the percentage of neutrophils ingesting 2 or more zymosan particles ex vivo

SECONDARY OUTCOMES:
neutrophil phagocytic capacity on alternate study days | 0 - 9 days
  Measured on alternate days and also as 'area under the curve' over the study period
Other measures of neutrophil function | 0-9 days
  May include but not limited to: ROS generation, migration capacity and apoptotic rate
Monocyte HLA-DR expression | 0-9 days
  Alternate days by flow-cytometry
Serum measures of inflammatory response | 0-9 days
  May include but not limited to: cytokine levels
Sequential organ failure assessment (SOFA) | up to end of study participation, a maximum of 30 days for each participant
Length of ICU stay | Up to end of participation in study, a maximum of 30 days
Incidence of ICUAIs (Intensive care unit acquired infection) | Up to end of study participation, a maximum of 30 days for each patients
  As defined by hospitals in europe link for infection control surveillance (HELICS)
All cause mortality | 30 days post randomisation
Number of days of mechanical ventilation | Up to end of study participation, a maximum of 30 days
Blood sample analysis | 0-9 days
  To measure safety of study medication from blood samples, which will include measures of Full blood count, white cell count (including differential), U&Es and LFTs, development of neutralising antibodies to GMCSF

CONTACTS AND LOCATIONS:
Overall Officials: John Simpson, Principal Investigator — Newcastle University
Locations (4):
- United Kingdom (4):
  - Queen Elizabeth Hospital, Gateshead, Tyne and Wear
  - Royal Victoria Infirmary, Newcastle upon Tyne, Tyne and Wear
  - Freeman Hospital, Newcastle upon Tyne, Tyne and Wear
  - Sunderland Royal Hospital, Sunderland